CLINICAL TRIAL: NCT03661619
Title: Tuberosity Versus Palatal Donor Site for Subepithelial Connective Tissue Graft in Root Coverage Therapy: a Randomized Clinical Trial (TOPGRAFT)
Brief Title: Tuberosity Versus Palatal Donor Site for Subepithelial Connective Tissue Graft in Root Coverage Therapy (TOPGRAFT)
Acronym: TOPGRAFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K171206J
Record Dates: First submitted 2018-06-15; First posted 2018-09-07 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-06

CONDITIONS: Gingival Recession
Keywords: Gingival recession; Root coverage; Periodontal plastic surgery; Subepithelial connective tissue graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Envelope technique + sub-epithelial connective tissue graft harvested from the palatal for root coverage procedure
  Interventions: Procedure: Sub-epithelial connective tissue graft harvested from the palatal for root coverage procedure
- Test Group (Experimental): Envelope technique + sub-epithelial connective tissue graft harvested from the tuberosity for root coverage procedure
  Interventions: Procedure: Sub-epithelial connective tissue graft harvested from the tuberosity for root coverage procedure

INTERVENTIONS:
Procedure: Sub-epithelial connective tissue graft harvested from the palatal for root coverage procedure — Envelope technique + sub-epithelial connective tissue graft harvested from the palatal for root coverage procedure
  Other Names: Palatal graft
  Arms: Control Group
Procedure: Sub-epithelial connective tissue graft harvested from the tuberosity for root coverage procedure — Envelope technique + sub-epithelial connective tissue graft harvested from the tuberosity for root coverage procedure
  Other Names: Tuberosity graft
  Arms: Test Group

SUMMARY:
Gingival recessions are characterized by the apical migration of the marginal gingivae toward the cemento-enamel junction. Our team in France reported that 84,6% of the population exhibited gingival recession. Other epidemiologic data report that 25% of an american population exhibit recessions deeper than 3mm.

Recessions may be associated with thermic or mecanic related pains and increased wear of the roots. It may causes aesthetic prejudice on smiling. It may also complicate prosthetic reconstruction when the volume of tissue are insufficient. A study on a Brazilian population reported that recessions negatively impacted the quality of life in terms of esthetics and root sensitivity.

Many surgical procedures have been created to treat these recessions. Most of them include a gingival graft by mean of a sub-epithelial connective tissue graft. Usually it is harvested in the hard palate. However, the early healing of the palate may be associated with important pain and discomfort. Another harvesting site is the retromolar tuberosity. It seems to be of higher tissular quality and lower healing complications. However its limited volume prevent the harvesting of large graft.

Almost no studies have compared the clinical outcome between palatal and tuberosity graft. A retrospective study of our team reported higher rate of complet root coverage with tuberosity graft versus palatal graft (OR=3,78 IC95%). After this observational study, our work introduce a interventional comparison between the two harvesting sites.

DETAILED DESCRIPTION:
Recruitment and inclusion:

Patients will be recruited from the consultation of the service of periodontology at Rothschild hospital, Paris, France. All eligible willing participant is included between 2 to 8 weeks before intervention. At that time, data are collected, including periodontal parameters and standardized photographs.

Randomization:

It is performed right before intervention by the operator via CleanWEB. Surgical protocol Both test and control groups will be treated with the same flap design. Patient will receive local anaesthesia at the recession and donor site (articaine hydrochloride 7200 mg/1.8 ml, adrenalin 1800 mcg/1.8 ml).

Envelope technique:

By means of a blade (Bard-Parker 15C; Beckton Dickinson) incision stars in the sulcus of the treated teeth, as tissue thickness permits, sharp dissection is used to form a partial-thickness supraperiosteal envelope extending 3 fo 5 mm internally and apically to areas of recession, undermining intermediate papillae. The supra-periosteal dissection will extend well into the mucosal tissues in order to gain flap mobility. The adjacent papillary tissues will be carefully detached by a full-thickness preparation in their buccal aspect, thus to allow for a coronal displacement of the mobilized buccal soft tissue complex.

In accord with the randomization process, one of the following techniques could be employed.

The donor area in the palate anesthetized by block anesthesia of the grater palatine and nasopalatine nerves with a local anesthetic agent containing epinephrine.

Palate : Single-incision technique In this technique, only a single incision parallel 2mm from the gingival margin is use to access to the donor site for graft harvesting. The angle of the blade is 90 degrees to the bone. After the first incision the blade is angle to approximately 135 degrees, and an undermining preparation toward the median is started within the first incision. With each new movement of the scalpel along the incision line, the angle is further flattened until the blade reaches a nearly parallel position to the bone surface. No vertical incisions are to be made, the goal of this procedure is to create a partial-thickness mucosal flap with a uniform thickness of 1 to 1.5 mm depending in the needs for the recipient site. The underlying CTG is separated from the surrounding connective tissue by making incisions to bone on the mesial, distal sides of the graft. The graft can then be removed by detaching it from the bony surface with a periosteal elevator. Suture of the donor site: crossed and parallel horizontal suspension sutures secure the incision and the donor site.

Tuberosity : Distal wedge technique The procedure starts with two converging incisions perpendicular to the tissue surface and 1.0-1.5 mm deep as far distal to the last molar as possible while remaining within the masticatory mucosa. Then, an undermining partial-thickness incision buccal and palatal up to the mesial surface of the last molar is made. The scalpel is guided successively parallel to the buccal or palatal soft tissue surfaces to yield a partial-thickness flap of uniform thickness throughout. After a supraperiosteal incision is made the wedge-shaped graft is removed from he donor site by sharp dissection. The covering epithelium on the upper part of the graft is consequently removed extraorally. The donor site is closed with an external horizontal mattress suture anchored to the periosteum. Additional single interrupted sutures can be used to completely close the wound.

Graft considerations Care should be taken to avoid graft dehydration from the moment when the graft is taken until the wound from the donor site is closed, so it should be store in a gauze soaked in physiologic saline until further use.

Extra oral modifications in SCTGs is often necessary, a fresh scalpel blade could be used to cut the graft to the desired size and shape and to thin the SCTG as needed, also fat and glandular tissue remnants detected on the graft should be removed.

Graft positioning and suturing The connective tissue graft is place in the created envelope, small parts of the CTG could be left uncovered when necessary to achieve a harmonious line of the gingival margin.

Prior to suturing, the contact points of the affected teeth need to be temporarily splinted with a flowable, light-curing resin material.

Suturing material is a non resorbable suture (Prolène 5.0: Ethicon - Cornelia, Georgia, USA).

Starting at the buccal aspect, the needle is guided through the buccal soft tissue complex approximately 5 mm apical to the tip of the papilla. so the needle will reappear in the base of the palatal papilla area. Consecutively, the needle will be wrapped around the splinted contact region and slid underneath the contact point to re-appear at the palatal side again without pinching any soft tissue. The same procedure is repeated once again, now starting from the palatal aspect.

Thereon the needle will be led over and placed underneath the contact point to re-appear at the buccal aspect again without pinching any soft tissue

Post-surgical protocol Patients have to avoid mechanical trauma or tooth brushing in the surgical sites for two weeks. Chlorhexidine rises are prescribed three times per day for two weeks. Two weeks after the surgery patients are instructed to mechanical tooth cleaning with a soft brush.

Following this, regular tooth brushing habits are resumed and chlorhexidine rinses discontinued.

Standardized photograph are also performed.

Follow up visit Supportive care are provided at 6 and 12 months. Data including periodontal parameters and standardized photographs are collected at the 6 months visit and at the12 months visit by an investigator different from the operator.

This is the last visit of the study. Further supportive care are normally provided at the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females must be at least 18 years of age.
2. Patients must be in good general health without any systemic diseases.
3. Presence of buccal gingival recession (Miller's Class I and II) >2 mm.
4. Identifiable cemento-enamel junction.
5. The tooth with a gingival recession is a vital tooth.
6. Accessible tuberosity.
7. Plaque Index and Gingival bleeding index less than 20%.
8. Use an atraumatic dental brushing technique.
9. Provide signed and dated informed consent form.
10. Social health insurance.

Exclusion Criteria:

1. The tooth with a gingival recession is a molar
2. Prosthetic crown, restoration or tooth decay involving the CEJ
3. Previous periodontal plastic surgery in the area
4. Smokers up to 10 per day.
5. Patient with untreated periodontal disease.
6. Presence of clinical signs of active periodontal disease
7. Known pregnancy in progress
8. Contraindication to surgery
9. Patient deprived of liberty or under legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Gingival recession | 12 months
  The distance from CEJ to the gingival margin in the mid-buccal site of the treated tooth. Recession will be measured where there is the greatest distance between the marginal gingiva and the cemento-enamel junction (CEJ) in the vertical direction.

SECONDARY OUTCOMES:
Pocket depth | 12 months
  on the mesio-, mid-, and disto-buccal sites, the distance from gingival margin to the bottom of the gingival sulcus.
Keratinized tissue heigth | 12 months
  The distance between the soft tissue margin and the mucogingival junction at the facial aspect of the tooth.
Aesthetic evaluation | 12 months
  A before-after scoring panel system will be used. Each preoperative and postoperative photograph is reframed for matching with a photo editing application and imported in presentation software.
  The views will be rated in one session by an independent professional examiner (periodontist).
  The observer will be masked to the patient, the operator, and the given treatment. The cosmetic results will be scored using the following five-point ordinal improvement scale:
  poor (1), fair (2), good (3), very good (4), and excellent (5).
  The observer will be asked to score for each before/after picture in eight parameters:
  1. -Global esthetic appearance
  2. -Degree of root coverage
  3. -Color match
  4. -Texture match
  5. -Volume match
  6. -Lack of hypertrophic scars
  7. -Existing keratinized tissues
  8. -Gingival contour
Post operative morbidity assessment | 2 weeks
  Each patient will answer a questionnaire. Post operative morbidity will be evaluated at 2 weeks regarding the intensity of the given event and be marked on a 10 points visual analogue scale (VAS).
Aesthetics and satisfaction assessment | 12 months
  Aesthetics and satisfaction will be evaluated at the 12-months follow-up visit. Patients will be asked to select among 3 items.
Duration of surgery | intraoperative
  How long in minutes last the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BOUCHARD, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No